CLINICAL TRIAL: NCT02220829
Title: Prophylactic Versus Therapeutic Alpha-Blockers in Prostate Cancer Patients Undergoing Radical Course Radiation Therapy ± HDR Boost. a GROUQ Phase III Randomized Clinical Trial (PCS-VII).
Brief Title: Comparative Study of Use of Alpha-Blockers to Treat Symptoms in Prostate Cancer Patients Undergoing Radiation Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sir Mortimer B. Davis - Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Dr. Tamim Niazi, Radiation Oncologist, Sir Mortimer B. Davis - Jewish General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PCS VII
Record Dates: First submitted 2014-08-18; First posted 2014-08-20 (Estimated); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Urinary Problems; Prostate Cancer
Keywords: alpha-blocker; symptomatic urinary problems; radiation therapy; prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — silodosin; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | US Export: No

ARMS (2):
- Preventive administration of Rapaflo (Active Comparator): Rapaflo treatment will start on day one of radiation therapy (early administration- before symptoms onset) and continue for a total duration of 6 months: 8 mg daily during 4 months and 8 mg every other day for 2 months.
  Interventions: Drug: Preventive administration of Rapaflo
- Standard care (Other): Administration of alpha-blocker Rapaflo at the onset of symptomatic urinary problems caused by radiation therapy. 8 mg of Rapaflo is administered daily until disappearance of symptoms.
  Interventions: Drug: Standard Care

INTERVENTIONS:
Drug: Preventive administration of Rapaflo — Rapaflo treatment: 8 mg daily during 4 months and 8 mg every other day for 2 months.
  Other Names: Rapaflo; Silodosin
  Arms: Preventive administration of Rapaflo
Drug: Standard Care — Administration of alpha-blocker Rapaflo only at onset of symptoms.
  Other Names: Rapaflo; Silodosin
  Arms: Standard care

SUMMARY:
Approximately 50%-95% of prostate cancer patients undergoing radiation therapy (RT) develop symptomatic urinary problems .These symptoms can significantly diminish a patient's quality of life during and shortly after therapy. Alpha1-blockers, such as Rapaflo, act to decrease resistance to urinary flow.

This multi-institutional phase III trial is designed to compare standard of care versus preventive treatment with Rapaflo for prostate cancer patients, regardless of risk group, whose treatment consists of radical radiation therapy. We plan to recruit 188 patients across Quebec who will be randomized into two arms: rapaflo prescribed at start of radiation therapy or if/when symptoms appear.

DETAILED DESCRIPTION:
The efficacy of Rapaflo treatment will be assessed using the International Prostate Symptom Score (IPSS). The IPSS will be assessed at baseline before RT, 4 weeks into RT, the last day of RT, and monthly thereafter for a total duration of 6 months from start of RT. Patients will have 2 more IPSS assessments at 9 and 12 months. The total duration of follow-up will be one year from start of RT. We will compare the rate of IPSS increase in the Rapaflo group compared to the standard arm at different time point (4 weeks, 6 weeks and at the end of treatment). We will also determine the rate of IPSS return to baseline at 4 and 12 weeks after the end of treatment. The rate of therapy dependence in the 2 arms will be evaluated at 20 and 26 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adult male 18 years of age or older
* Patients with confirmed diagnosis of adenocarcinoma of the prostate.
* The primary treatment should be external beam radiation therapy (EBRT) with or without high dose rate (HDR) brachytherapy boost.
* Clinical or radiological diagnosis of T1a - T3b.
* No limitation with respect to Gleason score.
* No limitation with respect to total Prostate-specific Antigen (PSA) value.
* Karnofsky performance score (KPS) of ≥ 70.

Exclusion Criteria:

* Small cell cancer of the prostate
* T4 disease, invading bladder or rectum.
* Adjuvant or salvage radiation therapy
* Brachy monotherapy
* KPS < 70

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2023-04 (Actual); Study Completion 2023-08 (Actual)

PRIMARY OUTCOMES:
To determine the rate of increase and the mean difference from the baseline IPSS score in the alpha-blocker (Rapaflo) group compared to the standard arm. | IPSS will be assessed before radiation therapy (RT), 4 weeks into RT, the last day of RT, and monthly for first 6 months and also at 9 and 12 months from the start of RT.

SECONDARY OUTCOMES:
To determine the rate of IPSS return to baseline, in the alpha-blocker (Rapaflo) group compared to the standard after the end of radiation treatment. | IPSS score will be assessed at before radiation therapy (RT), at 4 and 12 weeks after the end of RT.
To determine the rate of therapy dependence in both groups. | At 3 and 6 months from start of radiation therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Tamim Niazi, MD, Principal Investigator — Jewish General Hospital, McGill University
Locations (1):
- Jewish General Hospital, McGill University, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pollack A, Zagars GK, Starkschall G, Childress CH, Kopplin S, Boyer AL, Rosen II. Conventional vs. conformal radiotherapy for prostate cancer: preliminary results of dosimetry and acute toxicity. Int J Radiat Oncol Biol Phys. 1996 Feb 1;34(3):555-64. doi: 10.1016/0360-3016(95)02103-5. PMID 8621278
- [Background] Tsumura H, Satoh T, Ishiyama H, Tabata K, Kotani S, Minamida S, Kimura M, Fujita T, Matsumoto K, Kitano M, Hayakawa K, Baba S. Comparison of prophylactic naftopidil, tamsulosin, and silodosin for 125I brachytherapy-induced lower urinary tract symptoms in patients with prostate cancer: randomized controlled trial. Int J Radiat Oncol Biol Phys. 2011 Nov 15;81(4):e385-92. doi: 10.1016/j.ijrobp.2011.04.026. Epub 2011 Jun 12. PMID 21664068